CLINICAL TRIAL: NCT00328965
Title: An Open Label, Multi-centre, Single Arm Phase IV Study to Evaluate the Antihypertensive Effect of Lacidipine in Mild to Moderate Essential Hypertension Patients With Type 2 Diabetes in Korea
Brief Title: Lacidipine In Mild To Moderate Essential Hypertension Patients With Type 2 Diabetes In Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAC103842; VAXAR FEV
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 2; Essential Hypertension
Keywords: Korean patients; Type 2 diabetes; Endothelial function; lacidipine; Essential hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Essential Hypertension | interventions — lacidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacidipine (Other): All subjects who meet eligiblity criteria receive 2mg for the first 4 weeks in an open manner. If target systolic blood pressure is not ahcieved, subject can increase the dose to 4mg and then 6mg consequently.
  Interventions: Drug: Lacidipine

INTERVENTIONS:
Drug: Lacidipine — Lacidipine 2, 4, 6mg

SUMMARY:
This study was designed to evaluate the anti-hypertensive efficacy of lacidipine in hypertensives with Type 2 diabetes and effectiveness on endothelial cell function in Korean population.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed as essential hypertension or not treated in the past 2 weeks(If the subject took medication in the past 2 weeks, a wash-out period of at least 2 weeks will be completed prior to performing screening (week -2) assessments)
* Mean seated SBP at screen visit = 130mmHg (as measured by a mercury sphygmomanometer)
* Type 2 diabetes (American Diabetes Association criteria 2004) and HbA1C <11%
* Agree to practice acceptable contraceptive measures during the study, and for 30 days after the last dose of study medication is taken if the subject a female of child-bearing potential
* Provide written informed consent

Exclusion criteria:

* Mean seated SBP of > 180 mmHg
* Known or suspected secondary hypertension
* Anemia defined by haemoglobin concentration < 10.0 g/dL
* Hemoglobinopathy or peripheral vascular disease
* Clinically significant renal or hepatic disease (i.e., subjects with serum creatinine = 2.0 mg/dL; Alanine aminotransferase, Aspartate aminotransferase, total bilirubin, or alkaline phosphatase > 2.5 times the upper limit of the normal reference range)
* Unstable or severe angina, coronary insufficiency, or any congestive heart failure requiring pharmacologic treatment
* Chronic disease requiring intermittent or chronic treatment with oral, intravenous, or intra-articular corticosteroids (i.e. only use of topical, inhaled or nasal corticosteroids is permissible)
* Female who is lactating, pregnant, or planning to become pregnant
* clinically significant abnormality identified at screening which in the judgement of the investigator makes the subject unsuitable for inclusion in the study (e.g. physical examination, laboratory tests, or electrocardiogram etc.)
* Acute or chronic metabolic acidosis or a history of diabetic ketoacidosis

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To investigate the clinical effectiveness of lacidipine on elevated systolic blood pressure (SBP) in Korean patients aged 35 to 75 years. | 12 weeks from baseline

SECONDARY OUTCOMES:
To investigate the clinical effectiveness of lacidipine on elevated diastolic blood pressure and endothelial function by flow-medicated vasodilation and measurement of markers of inflammation in Korean patients aged 35 to 75 years with type 2 diabetes. | 12 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, M.D., PH.D., Study Director — GlaxoSmithKline